CLINICAL TRIAL: NCT06704854
Title: Influence of Acute Daily Workload Changes on Low-frequency Fatigue Morning Scores Throughout an In-season Soccer Microcycle
Brief Title: Influence of Acute Daily Workload Changes on Low-frequency Fatigue Morning Scores
Status: Not yet recruiting | Type: Observational
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Other Study IDs: ST_Myo_weekly
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Fatigue Intensity
Keywords: fatigue; low-frequency fatigue; soccer
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Screening Platform — assessment of low-frequency fatigue using myocene
  Other Names: assessment of low-frequency fatigue

SUMMARY:
In recent years, the increased demands of both training and competition have heightened the need of load monitoring among soccer players. However, adopting metrics that comprehensively capture the intricacies of neuromuscular fatigue remains a challenge. Assessing low-frequency fatigue may contribute to fill this gap, as it provides an objective measure to evaluate muscle function readiness. Thus, the aim of this study was to examine whether variability in low-frequency fatigue morning scores are related to training external load acute changes throughout the in-season microcycle.

ELIGIBILITY:
Inclusion Criteria:

* elite soccer players

Exclusion Criteria:

* injured athletes

Ages: 16 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Elite soccer players competing at the highest national level
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2024-12-03 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
low-frequency fatigue | Day 1 (0 hours), Day 2 (24 hours), Day 3 (48 hours), Day 4 (72 hours), Day 5 (96 hours), Day 6 (120 hours)

IPD SHARING:
Plan to Share IPD: Undecided